CLINICAL TRIAL: NCT04867577
Title: Investigation on Cement Leakage on Vertebroplasty and Reconstruction for Spinal Compression Fracture
Brief Title: Assessement of Vertebroplasty-related Cement Leakage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202012233RIND
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Vertebral Fracture
Keywords: vertebra
MeSH Terms: conditions — Spinal Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- vertebral osteoporotic compression fracture: Patients with osteoporotic vertebral compression receiving vertebroplasty or cemented screws reconstruction
  Interventions: Diagnostic Test: CT scan of lung and spine

INTERVENTIONS:
Diagnostic Test: CT scan of lung and spine — Dual energy CT scan of thorax and spine

SUMMARY:
Vertebral compression fracture is a common disorder in elderly patients. Vertebroplasty or surgical fixation are therefore commonly performed, in which bone cement is injected and help to provide additional support for unstable fracture to ease the pain. Cement leakage to paraspinal vein is very common and often taken as indicator of endpoint of the procedure. However, the leaked cement entering venous system can go to right heart and cause pulmonary embolism sometimes. The prevalence and pattern of this problem is largely unknown, especially subclinical condition. In this project, we intend to perform in vivo investigation of the cement distribution under different injection conditions. We also plan to conduct a clinical study to investigate the pattern, prevalence, and risk factor of cement venous leakage and pulmonary embolism. The study is a prospective cohort design, in which we plan to recruit 60 patients who receive vertebroplasty or cemented pedicle screws fixation for vertebral compression fracture. Plain X ray and computed tomography (CT) will be performed after operation. For CT, plain CT for operated site and dual energy acquisition for pulmonary vasculature will be performed, in which the pulmonary perfusion will be detected precisely. The different modalities can help delineate of radiological pattern of cement leakage. Spine surgeon, interventional radiologist, neuroradiologist, and thoracic radiologist will participate in this project. Experience on the optimal technique for cement use under fluoroscope is expected. The knowledge obtained in this study can be used in clinical ground and translate into academic outcome and clinical patient care.

DETAILED DESCRIPTION:
Background Vertebral compression fracture is a common disease. Most of them are osteoporotic and minority of them are pathological. It cause severe pain and compression to neuronal tissue, leading to debilitating symptom and deficits. The quality of life can be reduced; long-term bed ridden can also cause morbidity and mortality. It is thus a major public health issue. Vertebroplasty and related procedure is an invasive procedure to restore vertebral stability by injection bone cement, usually under minimal percutaneous approach. Because of its immediate efficacy of pain relief, it is very popular and common procedure.

However, the cement is liquid before it become solid in the vertebrae. It can spread into venous system sometime, and even going into pulmonary circulation system. The latter cause pulmonary thromboembolism. Operators usually try their best to avoid such complication. Practically, severe complication is rare. According to prior literature, the cement leakage range from 2.1 to 26%. It indicate the problem is actually common. On the other hand, the cement can not be lysed by usual anticoagulant treatment. Detection of this condition can be of clinical importance.

Currently, the clinical epidemiology of cement leakage after vertebroplasty is not well studied. Many factors can contribute its occurrence, including technical, material, and patient-specific reasons. Although operators have their approach to avoid such conditions, there are little evidence to support the efficacy of individual preventive method. Actually, some operator tolerate minor paraspinal leakage because they believe it can achieve optimal cement filling in the vertebrae. However, it is unclear the relationship between paraspinal leakage and pulmonary embolism.

In detection of pulmonary thromboembolism, imaging method is mainstream. Currently, dual energy CT scan can provide optimal diagnosis of leaked cement and pulmonary perfusion status. The iodine map derived from material decomposition provide an easy way to detect perfusion defect. It can be used to detect and classify cement pulmonary embolism.

In this study, we aim to evaluate the clinical epidemiology of cement leakage in vertebroplasty and related surgery, focusing on the prevalence, severity, and risk factors. Based on the reference dual energy CT, we also want to investigate its imaging characteristics.

Study designs This is a prospectively hospital-based cohort study. We tend to enroll 60 patients in one year, in whom receive vertebroplasty or cemented screws for osteoporotic-related vertebral compression fracture. The postoperative spinal and thoracic imaging will be used to detect paraspinal and pulmonary embolism.

Inclusion citieria

1. Age > 20 years
2. Osteoporotic vertebral compression fracture, receiving vertebroplasty o cemented screws fixation

Exclusion criteria

1. Active infection,
2. Rapid neurological deterioration,
3. Bleeding tendency
4. Impaired renal function (serum creating > 1.5mg/dL)
5. Severe allergic reaction to contrast medium
6. Pregnant or breast-feeding women

Operation and clinical follow-up The enrolled patient will receive plain radiograph before operation. After operation, the plain radiograph of thorax and spine will be performed after regain ambulation ability. The thoracic and vertebral CT scan will be performed within one month. The demongraphic data will be record. The surgical details, including methods, location, material used, cement amount and component, will be recorded. Any surgical complication within one month will be recorded.

Imaging method

1. Vertebral and thoracic plain radiograph, in routine method, before and after operation
2. Dual energy thoracic CT scan after operation Contrast medium injection to highlight pulmomary artery. Post-processing to form iodine map to detect perfusion defect. P
3. Spinal vertebral CT of surgical location after opeation

Statistical analysis Detailed imaging analysis to detect prevalence and severity of paraspinal and pulmonary cement leakage and embolism will be recorded. The imaging characteristics will be analysed.The demographic, surgical, and material factors will be analysed with imaging findings in details with common statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* vertebral compression fracture requiring vertebroplasty or cemented transpedicular screws fixation
* older than 20 year old

Exclusion Criteria:

* active infection
* progressive neurological deterioration,
* coagulopathy
* renal insufficiency (serum creatinine > 1.5 mg/dL
* severe allergic reaction to contrast medium
* pregnant or breast-feeding women

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with vertebral compression fracture requiring vertebroplasty or cemented transpedicular screws fixation
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-04-30 (Estimated); Primary Completion 2022-03-29 (Estimated); Study Completion 2022-03-29 (Estimated)

PRIMARY OUTCOMES:
prevalence of pulmonary embolism | 6 months
  detection of cement pulmonary embolism on contrast enhanced dual energy CT

SECONDARY OUTCOMES:
prevalence of paraspinal venous leakage | 6 months
  detection of paraspinal cement leakage on CT

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Heng Lin, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
IPD is provided under request to principal investigator